CLINICAL TRIAL: NCT04822610
Title: Comparison of Analgesic Effectiveness of Ultrasound Guided Interscalene Block Versus Suprascapular With Axillary Block in Shoulder Arthroplasties
Brief Title: Comparison of Interscalene Block and Suprascapular With Axillary Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principal Investigator, M.D., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/1562
Record Dates: First submitted 2021-01-19; First posted 2021-03-30 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Shoulder Arthroplasty; Ultrasound Guided
Keywords: axillary block; suprascapular block

STUDY DESIGN:
Intervention Model Description: Study group - Study group- Control group
Who Masked: Outcomes Assessor
Masking Description: open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group: interscalene block + IV PCA (Experimental): preop usg guided interscalene block and IV PCA
  Interventions: Procedure: interscalene block
- Study group: suprascapular block + axillary block + IV PCA (Experimental): preop usg guided suprascapular block + axillary block and IV PCA
  Interventions: Procedure: suprascapular block + axillary block
- Control group: IV PCA (No Intervention): no block + IV PCA

INTERVENTIONS:
Procedure: interscalene block — peripheral nerve block
  Arms: Study group: interscalene block + IV PCA
Procedure: suprascapular block + axillary block — peripheral nerve block
  Arms: Study group: suprascapular block + axillary block + IV PCA

SUMMARY:
In this study, the investigators are going to compare the analgesia effectiveness of interscalane block and suprascapular with axillary block in shoulder arthroplasties

DETAILED DESCRIPTION:
In the preoperative period, the participants will be taken to the block room. The participants will be monitored, standard sedation will be applied.

The first group will be get interscalene block. The second group will be get suprascapular and axillary block. The third group patient will be get no block. Afterwards, the participants will be operated under general anesthesia. A patient-controlled analgesia device will be attached to each group of participants and their postoperative follow-up will be made.

ELIGIBILITY:
Inclusion Criteria:

* accepting the study protocol,
* age older than 18 years and younger than 90 years,
* undergoing shoulder arthroplasty surgery
* the American Society of Anesthesiologist (ASA) physical status of I-II-III-IV

Exclusion Criteria:

* severe respiratory distress
* patients with local anesthetic allergy
* contralateral hemidiaphragmatic parrhesia
* recurrent laryngeal nerve palsy
* infection at the injection site
* coagulation disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Opioid (mg) consumption | 48 hours
  Opioid (mg) consumption
Measurement of postoperative pain | 48 hours
  VAS (visual analog scale) (0: no pain, 10: the worst pain imaginable)

OTHER OUTCOMES:
Operation time | during surgery
  minutes
Hospital stay | postoperative period up to 3 days
  days
Postoperatif complication | postoperative period up to 3 days
  yes-no
Patient satisfaction | postoperative period up to 3 days
  5-point Likert scale: very satisfied (= 5), relatively satisfied (= 4), fairly satisfied (= 3), relatively dissatisfied (= 2) and very dissatisfied (= 1)
Beck Depression Inventory (BDI) | Will be done 3 times 1- on pre-operative hospitalization 2- in the hospital after surgery 3- in the 1st month follow-up after surgery
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Ozkan, MD, Principal Investigator — Istanbul Unıversity, Istanbul Faculty of Medicine, Anesthesiology
Locations (1):
- Istanbul University, Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toma O, Persoons B, Pogatzki-Zahn E, Van de Velde M, Joshi GP; PROSPECT Working Group collaborators. PROSPECT guideline for rotator cuff repair surgery: systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2019 Oct;74(10):1320-1331. doi: 10.1111/anae.14796. Epub 2019 Aug 7. PMID 31392721
- [Background] Lee SM, Park SE, Nam YS, Han SH, Lee KJ, Kwon MJ, Ji JH, Choi SK, Park JS. Analgesic effectiveness of nerve block in shoulder arthroscopy: comparison between interscalene, suprascapular and axillary nerve blocks. Knee Surg Sports Traumatol Arthrosc. 2012 Dec;20(12):2573-8. doi: 10.1007/s00167-012-1950-5. Epub 2012 Mar 21. PMID 22434159
- [Background] Park JY, Bang JY, Oh KS. Blind suprascapular and axillary nerve block for post-operative pain in arthroscopic rotator cuff surgery. Knee Surg Sports Traumatol Arthrosc. 2016 Dec;24(12):3877-3883. doi: 10.1007/s00167-015-3902-3. Epub 2016 Jan 5. PMID 26733274
- [Background] Cho N, Kang RS, McCartney CJL, Pawa A, Costache I, Rose P, Abdallah FW. Analgesic benefits and clinical role of the posterior suprascapular nerve block in shoulder surgery: a systematic review, meta-analysis and trial sequential analysis. Anaesthesia. 2020 Mar;75(3):386-394. doi: 10.1111/anae.14858. Epub 2019 Oct 3. PMID 31583679